CLINICAL TRIAL: NCT00200876
Title: Neurochemical Mediation of Placebo Responses in Humans
Brief Title: Effects of Anticipation of Pain Relief on Brain Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jon-Kar Zubieta, Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: R01AT001415-01A1 (NIH); R01AT001415-01A1 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Pain
Keywords: Positron-Emission Tomography; Endorphins; Pain Relief; Opioid Receptors; Stress; Analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Hypertonic saline is a challenge to activate endogenous opioid systems as assessed with positron emission tomography. There is no treatment involved. Isotonic saline is the control.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pain challenge (Active Comparator)
  Interventions: Procedure: Hypertonic saline; Procedure: Isotonic saline
- non-painful control (Sham Comparator)
  Interventions: Procedure: Hypertonic saline; Procedure: Isotonic saline

INTERVENTIONS:
Procedure: Hypertonic saline — To elicit pain
Procedure: Isotonic saline — Non-painful control

SUMMARY:
This study will use brain imaging technology to examine chemical systems in the brain that suppress pain and stress when an individual has an expectation of pain relief.

DETAILED DESCRIPTION:
Evidence suggests that the expectation of pain relief, even if a person receives only a placebo, can provide actual therapeutic benefits. The µ-opioid receptor system, located in the brain, is activated during anticipation of pain relief; this activation suppresses stress and pain responses. This study will use brain imaging technology to examine the effects of a placebo intervention on µ-opioid neurotransmitters. Examination of the factors that regulate these placebo-activated neurotransmitter responses will clarify the overall neurobiology underlying variations in the responses to placebos, as well as pain and other stressful conditions, ultimately leading to the optimization of medical and psychological interventions.

This study will last several hours during one study visit. Participants will receive both a painful and a painless injection while undergoing positron emission tomography (PET) brain imaging. The painful injection will consist of small amounts of hypertoninc saline (concentrated saline that causes cell shrinkage) in the jaw muscle over a 20-minute period. Several minutes after participants receive hypertonic saline, they will receive an injection with isotonic saline not associated with pain in the opposite jaw muscle. After participants receive the injections, they will either be told or not be told about a pain relief intervention. PET imaging will continue as participants either anticipate or do not anticipate pain relief. Participants will be asked about their pain levels repeatedly throughout the study; their responses will be entered into a computer-controlled system which will modulate rates of saline infusion.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with all study requirements

Exclusion Criteria:

* Presence of pain at study entry
* Personal or first-degree (e.g., mother, father, sister, brother) family history of neurologic or psychiatric disorders
* History of substance abuse or dependence
* Left-handed or ambidextrous
* Positive urine toxicology screen
* Acute or uncorrected medical illness that may interfere with the study
* Unable to tolerate brain scanning procedures
* Current treatment with antipsychotics, mood stabilizers, isoniazid (a drug for tuberculosis [TB]), glucocorticoids/mineralocorticoids, psychostimulant appetite suppressants, or centrally active antihypertensive drugs
* Treatment with hormones, antidepressants, or opioids within 6 months prior to study entry
* Treatment with sedative hypnotic medications or over-the-counter sleeping aids within 1 month prior to study entry
* Diagnosis of depression
* Competitive exercise, or exercise exceeding 1 hour each day
* Regular smoking within 5 years prior to study entry

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2003-09; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Placebo-induced activation of brain opioid neurotransmission | 90 min

CONTACTS AND LOCATIONS:
Overall Officials: Jon-Kar Zubieta, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No